CLINICAL TRIAL: NCT03359213
Title: Phase II Study of JR-141 in Patients With Mucopolysaccharidosis II
Brief Title: A Study of JR-141 in Patients With Mucopolysaccharidosis II (BR21)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: JCR Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JR-141-BR21
Record Dates: First submitted 2017-11-17; First posted 2017-12-02 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Mucopolysaccharidosis II
MeSH Terms: conditions — Mucopolysaccharidosis II

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- JR-141 1.0 mg/kg/week (Experimental)
  Interventions: Drug: JR-141
- JR-141 2.0 mg/kg/week (Experimental)
  Interventions: Drug: JR-141
- JR-141 4.0 mg/kg/week (Experimental)
  Interventions: Drug: JR-141

INTERVENTIONS:
Drug: JR-141 — IV infusion (lyophilized powder), 1.0 mg/kg/week
  Arms: JR-141 1.0 mg/kg/week
Drug: JR-141 — IV infusion (lyophilized powder), 2.0 mg/kg/week
  Arms: JR-141 2.0 mg/kg/week
Drug: JR-141 — IV infusion (lyophilized powder), 4.0 mg/kg/week
  Arms: JR-141 4.0 mg/kg/week

SUMMARY:
A Phase II open-label, randomized, parallel group, 2 sites (Brazil), designed to evaluate the safety and efficacy of 3 doses of study drug for the treatment of the MPS II.

ELIGIBILITY:
Inclusion Criteria:

* Males with confirmed diagnosis of MPS II, based on deficient activity of IDS in leucocytes or fibroblasts and/or pathogenic mutations identified in the IDS gene (if enzyme diagnosis was in dried blood spots or plasma, molecular genetics confirmation is mandatory).
* One of the following age groups:

  1. 0 to 3 years and 11 months old (6 patients, 2 in each dose)
  2. 4 years to 7 years and 11 months old (6 patients, 2 in each dose)
  3. 8 years or older (6 patients, 2 in each dose)
* Capable of providing written consent by himself, unless the patient is under the age of 18 years at the time of informed consent process, or it is not possible to obtain consent from the patient himself due to his intellectual disabilities associated with MPS II.
* In the case of a patient who is under the age of 18 years or from whom it is not possible to obtain consent due to his intellectual disabilities associated with MSP II, he may be included if written consent can be provided by legal representative; however written consent should be obtained from the patient himself too, wherever possible.
* Naïve patients or patients who are receiving enzyme replacement therapy with idursulfase could be included if provided treatment has been stable in the last 6 months and agree to interrupt the treatment at least one week before the first study drug infusion, and agree in suspending this treatment for the duration of the trial.

Exclusion Criteria:

* Refusal to sign the informed consent form.
* Unable to perform the study procedures, except for neurocognitive testing.
* Previous engrafted BMT/HSCT.
* Surgical or other major medical intervention planned to occur before week 26.
* Participation in a clinical trial with an investigational drug in the last 12 months.
* Judged by the investigator or subinvestigator as being unable to undergo lumbar puncture, including those who have difficulties in taking a position for lumber puncture due to joint contracture or those who are likely to experience difficulty breathing during the lumbar puncture process.
* Judged by the investigator or subinvestigator to be ineligible to participate in the study due to a history of a serious drug allergy or sensitivity.
* Otherwise judged by the investigator or subinvestigator to be ineligible to participate in the study out of consideration for the subject safety.

Min Age: 0 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-07-26 (Actual); Primary Completion 2019-10-04 (Actual); Study Completion 2019-10-04 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events | 26 weeks
  * Adverse events
  * Antidrug antibodies
  * Blood pressures in mmHg
  * Heart rate in beats/minute
  * Respiratory rate in breaths/minute
  * Temperature in °C
  * Presence or absence of abnormalities for physical examination
  * Presence or absence of abnormalities for 12-lead electrocardiogram
  * Routine laboratory tests in blood (hematology, liver function, renal function, iron-related levels) and urine (urinalysis)

SECONDARY OUTCOMES:
Plasma Pharmacokinetic parameter [Maximum Plasma Concentration [Cmax]] | 21 hours after dosing at the first and last infusions
  Plasma concentration of JR-141
Plasma Pharmacokinetic parameter [Area Under the Curve [AUC]] | 21 hours after dosing at the first and last infusions
  Plasma concentration of JR-141
Liver and spleen volumes (MRI) | 26 weeks
Left ventricular mass by a standard 2-dimensional Doppler echocardiogram | 26 weeks
Urinary heparan sulfate concentrations | 26 weeks
Urinary dermatan sulfate concentrations | 26 weeks
Serum heparan sulfate concentrations | 26 weeks
Serum dermatan sulfate concentrations | 26 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Grupo de Pesquisa Clínica em Genética Médica - HCPA, Porto Alegre
  - Igeim - Unifesp, São Paulo

IPD SHARING:
Plan to Share IPD: No